CLINICAL TRIAL: NCT02729779
Title: Effectiveness of the Pilates Method Versus Aerobic Exercises in the Treatment of Chronic Non-specific Low Back Pain in the Elderly: Randomized Controlled Trial
Brief Title: Effectiveness of the Pilates Method Versus Aerobic Exercises in Elderly With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, PhD, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53162216.9.0000.0064
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (Experimental): Elderly will be submitted to a specific exercise program of modified Pilates method performed in the mat and apparatus. In the first session, participants will receive basic guidance on the Pilates training and activation of the power house. The session will be divided in: global warming and stretching (5 minutes), Pilates exercises for upper and lower limbs, abdomen and spine (45 minutes), global stretching (5 minutes) and local relaxing massage (5 minutes).The session will consist of a minimum of 5 exercises and a maximum of 15 Pilates exercises. The elderly will receive 16 individual sessions with duration of 60 minutes, twice a week, with a total of eight weeks of treatment.
  Interventions: Other: Pilates Group
- Aerobic Group (Active Comparator): The Aerobic Group will be submitted to an exercise program with global stretching (for lower and upper limbs and column with two repetitions and 30 seconds of maintenance in each segment) for 10 minutes, walking on a treadmill for 20 to 40 minutes and relaxing massage for 5 minutes. The intensity of the effort during walking on a treadmill will be based on a combination of heart rate (based on the percentage of maximum heart rate: 208 - (0.7 x age)) and rate of perceived effort assessed by the Borg scale. Exercise will be performed respecting the fraction of 50-75% of maximum heart rate and levels between 12 to 13 (moderate intensity) of the Borg scale. The elderly will receive 16 individual sessions with duration of 60 minutes, twice a week, with a total of eight weeks of treatment.
  Interventions: Other: Aerobic Group

INTERVENTIONS:
Other: Pilates Group — Elderly will be submitted to a specific exercise program of modified Pilates method performed in the mat and apparatus. In the first session, participants will receive basic guidance on the Pilates training and activation of the power house. The session will be divided in: global warming and stretching (5 minutes), Pilates exercises for upper and lower limbs, abdomen and spine (45 minutes), global stretching (5 minutes) and local relaxing massage (5 minutes).The session will consist of a minimum of 5 exercises and a maximum of 15 Pilates exercises. The elderly will receive 16 individual sessions with duration of 60 minutes, twice a week, with a total of eight weeks of treatment.
  Arms: Pilates Group
Other: Aerobic Group — Elderly will be submitted to an exercise program with global stretching (for lower and upper limbs and column with two repetitions and 30 seconds of maintenance in each segment) for 10 minutes, walking on a treadmill for 20 to 40 minutes, and relaxing massage for 5 minutes. The intensity of the effort during walking on a treadmill will be based on a combination of heart rate (based on the percentage of maximum heart rate: 208 - (0.7 x age)) and rate of perceived effort assessed by the Borg scale. Exercise will be performed respecting the fraction of 50-75% of maximum heart rate and levels between 12 to 13 (moderate intensity) of the Borg scale. The elderly will receive 16 individual sessions with duration of 60 minutes, twice a week, with a total of eight weeks of treatment.
  Arms: Aerobic Group

SUMMARY:
Chronic low back pain is potentially disabling for the elderly, and physical exercises are considered the best treatment for this problem. The Pilates method has been proven effective in the improvement of pain and function in patients with low back pain. However, the evidence about the effectiveness of Pilates method in the treatment of elderly patients with low back pain is scarce. Thus, the aim of this study is to investigate the effectiveness of the Pilates method compared to aerobic exercise in elderly with chronic non-specific low back pain. This randomized controlled trial with two arms and blinded assessor will include 74 patients aged between 65 and 85 years, of both sexes, complaining of chronic non-specific low back pain persisting for more than three months and pain intensity greater than 3 points in the Pain Numerical Rating Scale. The elderly will be randomized into two groups: Pilates Group (n = 37) with exercises based on Pilates method; and Aerobic Group (n = 37) with aerobic exercises, stretching and relaxation. Both groups will hold treatment twice a week with duration of 60 minutes for eight weeks. The primary outcomes will be: pain intensity and general disability assessed eight weeks after randomization. Secondary outcomes will be: pain intensity and general disability evaluated six months after randomization; global impression of improvement, specific disability and dynamic balance, muscle strength of the gluteus maximus, gluteus medius and lateral hip rotators and pressure pain threshold evaluated eight weeks and six months after randomization. We expect that the results of this study contribute to the clinical decision-making with respect to pain reduction and, consequently, improving balance and functionality of elderly with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Elderly complaining of non-specific low back pain for more than three months
* Pain intensity equal to or more than 3 points evaluated by the Pain Numerical Rating Scale in the last seven days.

Exclusion Criteria:

* Contraindication to physical exercise;
* Back with severe disease (fractures, tumors, inflammatory diseases, ankylosing spondylitis and nerve root compromise confirmed by neurological tests);
* Previous or scheduled back surgery ;
* Severe cardiorespiratory disease;
* Cancer;
* Cognitive impairment;
* Dependent gait;
* Patients who underwent physical therapy for low back pain in the last six months;
* Regular physical activity practitioners.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Eight weeks after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Disabitity | Eight weeks after randomization
  Disability associated with low back pain will be measured using the 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Pain intensity | Six months after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Disability | Six months after randomization
  Disability associated with low back pain will be measured using the 24-item Roland Morris Disability Questionnaire
Global impression of improvement | Eight weeks and six months after randomization
  Global impression of improvement will be measured by an 11-point Global Perceived Effect Scale
Specific disability | Eight weeks and six months after randomization
  Specific disability will be evaluated by an 11-point Patient-specific Functional Scale
Dynamic balance | Eight weeks and six months after randomization
  Dynamic balance will be evaluated by the 10-meter Walk Test (fast and normal speed)
Dynamic Balance | Eight weeks and six months after randomization
  Dynamic balance will be evaluated by the Sit-up Test
Muscle strength of the gluteus maximus, gluteus medius and lateral hip rotators | Eight weeks and six months after randomization
  Muscle strength will be evaluated by dynamometer
Pressure pain threshold | Eight weeks and six months after randomization
  Pressure pain threshold will be evaluated by digital pressure algometer

CONTACTS AND LOCATIONS:
Overall Officials: Cristina MN Cabral, PhD, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Oliveira NTB, Ricci NA, Dos Santos Franco YR, Salvador EMES, Almeida ICB, Cabral CMN. Effectiveness of the Pilates method versus aerobic exercises in the treatment of older adults with chronic low back pain: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2019 May 24;20(1):250. doi: 10.1186/s12891-019-2642-9. PMID 31122227